CLINICAL TRIAL: NCT00880932
Title: The Effect of Customized Alerts Versus Generic Alerts for the Prescription of Warfarin and NSAID
Brief Title: Warfarin and Non-Steroidal Anti-Inflammatory Drugs (NSAID) Customized Alert
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: UPenn School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 803787
Record Dates: First submitted 2009-04-13; First posted 2009-04-14 (Estimated); Last update posted 2009-04-14 (Estimated); Status verified 2009-04

CONDITIONS: Warfarin and NSAID
Keywords: warfarin; NSAID; The condition is the concomitant prescription of

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- customized electronic alert (Experimental): This intervention was not targeted to patients with a disease but to the providers. The intervention was not a drug but a customized electronic alert, requesting the prescriber to specify a "reason for override" whenever the combination drugs of warfarin and NSAID were ordered together.
  Interventions: Behavioral: Electronic Alert
- Standard practice (No Intervention): The control group was not patients but the providers. Providers in the control group continued with the standard practice of receiving passive alerts in the form of message boxes warning the provider not to prescribe the combination drugs warfarin and NSAID.

INTERVENTIONS:
Behavioral: Electronic Alert
  Arms: customized electronic alert

SUMMARY:
The hypothesis is that a newly formatted electronic alert that requires the prescriber to pause and enter a specific "reason for override" on this alert, will cause prescribers in the intervention group to be significantly less likely to prescribe the combination of warfarin and NSAID than prescribers in the control group.

ELIGIBILITY:
Inclusion Criteria:

* All resident physicians (RP) and nurse practitioners (NP) involved in inpatient care at two hospitals of the University of Pennsylvania

Exclusion Criteria:

* None

Sex: All
Age Groups: Child, Adult, Older Adult
Enrollment: 1865 (Actual)
Dates: Start 2006-08; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Decreased rate of prescription of the combination of warfarin and NSAID | 17 months

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital of the University of Pennsylvania and Penn Presbyterian Medical Center, Philadelphia, Pennsylvania, United States